CLINICAL TRIAL: NCT06962865
Title: A Randomized, Open, Controlled, Multicenter Phase II Clinical Study of RC108 in Combination With Furmonertinib Versus Furmonertinib for the First-Line Treatment of EGFR-Mutated Combined MET-Positive Unresectable Locally Advanced or Recurrent Metastatic NSCLC
Brief Title: A Phase Ⅱ Study of RC108 in Combination With Furmonertinib for the First-line Treatment of EGFR-Mutated Combined MET-Positive Unresectable Locally Advanced or Recurrent Metastatic NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC108-C006
Record Dates: First submitted 2025-04-30; First posted 2025-05-08 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-04

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Injections; aflutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): 1L, EGFR-Mutated Combined MET-Positive Unresectable Locally Advanced or Recurrent Metastatic NSCLC
  Interventions: Drug: RC108; Drug: Furmonertinib Mesilate Tablets Monotherapy
- Arm 2 (Active Comparator): 1L, EGFR-Mutated Combined MET-Positive Unresectable Locally Advanced or Recurrent Metastatic NSCLC
  Interventions: Drug: Furmonertinib Mesilate Tablets Monotherapy

INTERVENTIONS:
Drug: RC108 — RC108 in Combination With Furmonertinib
  Other Names: RC108 For Injection；
  Arms: Arm 1
Drug: Furmonertinib Mesilate Tablets Monotherapy — Furmonertinib
  Other Names: Furmonertinib

SUMMARY:
Evaluate the efficacy and safety of RC108 in combination with Furmonertinib against Furmonertinib for treatment of EGFR mutation combined with MET-positive unresectable locally advanced or recurrent metastatic NSCLC

DETAILED DESCRIPTION:
Primary objective: Evaluate the efficacy and safety of RC108 in combination with Furmonertinib against Furmonertinib for treatment of EGFR mutation combined with MET-positive unresectable locally advanced or recurrent metastatic NSCLC Secondary objective: Evaluate the pharmacokinetic and immunogenicity characteristics of RC108 in combination with Furmonertinib

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in the study and signed the ICF;
2. Male or female, aged 18-75 years;
3. All participants to be enrolled must be diagnosed with histopathologically or cytologically confirmed, unresectable locally advanced (stage IIIB/IIIC )or recurrent metastatic NSCLC (stage IV ) and not amendable to curative surgery or radiation as assessed by investigator;
4. For previously locally advanced or recurrent metastatic disease not treated with systemic antitumor therapy;
5. Carring 1 of 2 common EGFR mutations clearly associated with EGFR-TKI sensitivity (i.e., exon 19 deletion or L858R) and MET positivity;
6. Ability to provide at least 6 sections of tumor tissue specimens for staining and testing；
7. ECOG PS score 0 or 1；
8. At least one measurable lesion according to RECIST v1.1 criteria；
9. Expected survival ≥ 12 weeks;
10. Adequate bone marrow and organ function；
11. Female subjects of childbearing potential or male subjects whose partners are of childbearing potential must agree to use effective contraception from the time of signing the informed consent form until 6 months after the last dose, during which time the female subject is not breastfeeding and the male subject avoids sperm donation.

Exclusion Criteria:

1. Subjects with the presence of meningeal metastases, spinal cord compression, or active brain metastases；
2. Received ADC or MET inhibitors；
3. Suffering from refractory nausea and vomiting, chronic gastrointestinal disorders, inability to swallow pharmaceutical preparations, or previous major bowel resection that may prevent adequate absorption, distribution, metabolism, or excretion of oral medications;
4. Subjects with uncontrolled tumor-related pain；
5. Use of an investigational drug or major surgery within 4 weeks before the first dose;
6. Received any live vaccine within 28 days prior to the first dose or plan to be vaccinated during the study;
7. Subjects with uncontrolled or severe cardiovascular disease;
8. Presence of clinically uncontrollable third interstitial effusion;
9. Presence of severe lung disease, including but not limited to active tuberculosis, interstitial lung disease requiring treatment, radiation pneumonitis, etc.
10. Toxicity due to prior antineoplastic therapy has not recovered to National Cancer Institute Commonly Used Criteria Terminology for Generic Adverse Events, Version 5.0, Grade 0-1;
11. Persistent grade ≥2 sensory or motor neuropathy;
12. Active infections requiring systemic IV antibiotic therapy within 7 days before the first dose, allowing routine antimicrobial prophylaxis;
13. Positive test result for Human Immunodeficiency Virus (HIV) or history of Acquired Immune Deficiency Syndrome (AIDS);
14. Active hepatitis B or HCV-positive subjects;
15. Received systemic corticosteroid therapy with >10 mg/day prednisone or other immunosuppressive medications within 2 weeks before randomization;
16. Other malignant tumor within 5 years before signed the informed consent form;
17. Known hypersensitivity or delayed hypersensitivity to RC108, certain components of Furmonertinib or similar drugs or any contraindication to the drug;
18. Poor compliance and unable to complete the study procedures as assessed by investigator;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 24 months
  Investigator-assessed ORR

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 24 months
  Investigator-assessed PFS
Disease Control Rate (DCR) | 24 months
  Investigator-assessed DCR
Duration of Response (DoR) | 24 months
  Investigator-assessed DoR
Overall survival (OS) | 45 months
  Investigator-assessed OS
Number of participants with adverse events (AEs) | 24 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Incidence of RC108 anti-drug antibody (ADA) | 24 months
  Incidence, occurrence time and ADA titer of positive RC108 ADA and neutralizing antibodies
Pharmacokinetic profile of RC108 | 24 months
  Peak and trough concentrations of RC108 total antibody (TAb), conjugated antibody (ADC), free MMAE

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Zhang, Study Director — Hunan Cancer Hospital
Locations (34):
- China (34):
  - Beijing Chest Hospital,Capital Medical Unniversity, Beijing
  - The Fifth Medical Center of Chinese People's Liberation Army General Hospital, Beijing
  - Binzhou Medical University Hospital, Binzhou
  - Jilin Cancer Hospital, Changchun
  - The Second Xiangya Hospital Of Central South University, Changsha
  - Changzhou Cancer Hospital, Changzhou
  - Sichuan Cancer Hospital, Chengdu
  - West China hospitial of SiChuan University, Chengdu
  - Chongqing University Cancer Hospitai, Chongqing
  - Fujian Cancer Hospital, Fuzhou
  - Ganzhou cancer Hospitial, Ganzhou
  - Affiliated Cancer Hospital of Guangzhou Medical University, Guangzhou
  - The First Affiliated Hospital of Wenzhou Medical University, Guilin
  - The Second Affiliated Hospital of Guilin Medical University, Guilin
  - Sir Run Run Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Anhui Provincial cancer hospital, Hefei
  - The First hospitial of Anhui Medicine University, Hefei
  - Jinan Central Hospital, Jinan
  - Shandong Cancer Hospital, Jinan
  - The First hospitial of Lanzhou University, Lanzhou
  - Linyi People's Hospital, Linyi
  - THE FIRST HOSPITAI OF CHINA MEDICAL UNIVERSITY,No. 155, Nanjing North Street, Heping District, Shenyang City, Liaoning Province, Shenyang
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang
  - Shanxi Cancer Hospital, Taiyuan
  - Taizhou hospitial of Zhejiang province, Taizhou
  - Tianjin Chest Hospital, Tianjin
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Xiangyang Central Hospital, Xiangyang
  - The Second People's Hospital of Yibin City, Yibin
  - Yiyang Central Hospital, Yiyang
  - Yueyang Central Hospital, Yueyang
  - Yunnan Cancer Hospital, Yunnan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou